CLINICAL TRIAL: NCT07406932
Title: A Study on the Efficacy and Safety of JAK Inhibitors Versus Calcineurin Inhibitors as Initial Therapy for Interstitial Lung Disease Associated With Antisynthetase Syndrome
Acronym: JAKCNIASSILD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Qinghong Liu, Physician, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JAKCNIASSILD
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Antisynthetase Syndrome; Interstitial Lung Disease (ILD)
MeSH Terms: conditions — Antisynthetase syndrome; Lung Diseases, Interstitial | interventions — Janus Kinase Inhibitors; Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JAK inhibitor group (Experimental): Participants in this arm will receive one of the JAK inhibitors (tofacitinib 5 mg twice daily, or baricitinib 4 mg once daily, or upadacitinib 15 mg once daily) in combination with a standard glucocorticoid regimen (methylprednisolone 0.5g IV for 3 days, followed by oral prednisone 0.8-1.0 mg/kg/day tapered to 7.5 mg/day over 12 months). Treatment duration is 12 months.
  Interventions: Drug: JAK Inhibitor
- Calcineurin inhibitor group (Experimental): Participants in this arm will receive either tacrolimus (0.075 mg/kg/day in two divided doses) or cyclosporine (2-5 mg/kg/day in two divided doses) in combination with the same standard glucocorticoid regimen as the experimental group. Treatment duration is 12 months.
  Interventions: Drug: Calcineurin Inhibitors (CNI)

INTERVENTIONS:
Drug: JAK Inhibitor — Oral JAK inhibitors (tofacitinib 5 mg twice daily, or baricitinib 4 mg once daily, or upadacitinib 15 mg once daily) administered in combination with standard glucocorticoid therapy for 12 months.
  Arms: JAK inhibitor group
Drug: Calcineurin Inhibitors (CNI) — Oral calcineurin inhibitors (tacrolimus 0.075 mg/kg/day in two divided doses, or cyclosporine 2-5 mg/kg/day in two divided doses) administered in combination with standard glucocorticoid therapy for 12 months.
  Arms: Calcineurin inhibitor group

SUMMARY:
This study is a prospective investigation comparing the efficacy and safety of Janus kinase inhibitors versus calcineurin inhibitors as initial therapy for interstitial lung disease associated with antisynthetase syndrome. The goal is to determine which treatment is more effective at improving lung function and preventing disease progression, while comparing their safety profiles. The findings will help provide clearer treatment guidance for doctors and patients.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label, prospective study. Eligible adults with interstitial lung disease associated with antisynthetase syndrome (ASS-ILD) who are treatment-naïve will be randomly assigned to receive either a JAK inhibitor (tofacitinib 5 mg twice daily, or baricitinib 4 mg once daily, or upadacitinib 15 mg once daily) or a calcineurin inhibitor (tacrolimus 0.075 mg/kg/day in two divided doses, or cyclosporine 2-5 mg/kg/day in two divided doses), both in combination with a standard glucocorticoid regimen. The primary endpoint is the 12-month survival rate. Secondary endpoints include changes in lung function, high-resolution CT (HRCT) scores, glucocorticoid dosage reduction, and the proportion of patients achieving low disease activity. Safety and laboratory parameters will be closely monitored throughout the 12-month treatment and follow-up period. Statistical analyses will compare the efficacy and safety profiles between the two treatment arms, and subgroup analyses will be performed to explore potential predictors of treatment response.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to 75 years. Meet the 2017 EULAR/ACR diagnostic criteria for Anti-synthetase Syndrome (ASS). Presence of Interstitial Lung Disease (ILD) confirmed by High-Resolution Computed Tomography (HRCT).

Active disease requiring initiation or intensification of immunosuppressive therapy, with no prior use of glucocorticoids, immunosuppressants, or biologics.

Signed informed consent form.

Exclusion Criteria:

Diagnosis of Rapidly Progressive ILD (RP-ILD), defined as worsening dyspnea within 1 month and PaO2/FiO2 ratio < 250 mmHg.

Active uncontrolled severe infection, malignancy, or major organ failure. Pregnancy or lactation. Contraindications to the study drugs. Concurrent use of other immunosuppressants or biologics.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
12-month survival rate | 12 months
  Proportion of participants surviving at 12 months after randomization, with survival defined as the time from randomization to death from any cause.

SECONDARY OUTCOMES:
Annual decline rate of lung function (FVC% and DLCO%) | Change from baseline to 12 months
  The annual rate of decline in forced vital capacity (FVC% predicted) and diffusing capacity for carbon monoxide (DLCO% predicted), calculated as the change from baseline to 12 months.
Change in HRCT score | Change from baseline to 12 months
  Change in high-resolution computed tomography (HRCT) score from baseline to 12 months, assessed using a standardized scoring system.
Rate of glucocorticoid tapering | Over 12 months
  The rate of glucocorticoid dose reduction over 12 months, calculated as the time to achieve prednisone ≤7.5 mg/day or the cumulative glucocorticoid dose.
Proportion of patients achieving low disease activity (LDA) | At 6 months and 12 months
  Proportion of participants achieving low disease activity (LDA) at 6 and 12 months, defined as meeting all of the following criteria: no active arthritis without regular NSAID use; no active myositis with serum creatine kinase ≤ upper limit of normal; stable ILD with no decline in pulmonary function (FVC decline <5% and DLCO decline <10% in the past 6 months); no fever or other systemic manifestations with ESR <20 mm/h; stable glucocorticoid dose ≤7.5 mg/day (prednisone equivalent) for at least 3 months.